CLINICAL TRIAL: NCT06654570
Title: Effects of Vaginal Estrogen on Serum Estradiol During Aromatase Inhibitor Therapy in Breast Cancer Patients with Vulvovaginal Atrophy: a Prospective Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Johanna Mattson, Senior Medical Director, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001234-34
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: breast cancer, adjuvant, letrozole, estradiol, vulvovaginal atrophy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravaginal estradiol during adjuvant letrozole (Experimental): Eligible patients were treated with Vagifem® (17β-estradiol hemihydrate) 10 μg vaginal tablets for 12 weeks. Patients were instructed to insert one vaginal tablet daily using the provided applicator for 14 consecutive days, followed by one tablet twice weekly (Monday and Thursday evenings).
  Interventions: Drug: Intravaginal estrogen during adjuvant letrozole

INTERVENTIONS:
Drug: Intravaginal estrogen during adjuvant letrozole — Postmenopausal patients undergoing adjuvant letrozole therapy and experiencing VVA symptoms were treated with vaginal estradiol for 12 weeks. Gynecologic examination and symptom screening were conducted at baseline and after 12 weeks. Serum E2 levels were analyzed at baseline, and at two, four, eight, and 12 weeks. E2 levels were measured using both a routine liquid chromatography-tandem mass spectrometry (LC-MS/MS) method and a highly sensitive (hsE2-MS) LC-MS/MS method.

SUMMARY:
Purpose: This study aimed to analyze changes in serum estradiol (E2) levels during concurrent vaginal estradiol therapy and adjuvant letrozole in postmenopausal breast cancer (BC) patients with vulvovaginal atrophy (VVA). Secondary objectives included assessing the effects of therapy on vaginal atrophy, quality of life (QoL) and menopause-related symptoms.

Methods: Postmenopausal patients undergoing adjuvant letrozole therapy and experiencing VVA symptoms were treated with vaginal estradiol for 12 weeks. Gynecologic examination and symptom screening were conducted at baseline and after 12 weeks. Serum E2 levels were analyzed at baseline, and at two, four, eight, and 12 weeks. E2 levels were measured using both a routine liquid chromatography-tandem mass spectrometry (LC-MS/MS) method and a highly sensitive (hsE2-MS) LC-MS/MS method.

DETAILED DESCRIPTION:
The study was conducted between November 2020 and May 2024 at the Comprehensive Cancer Center, Helsinki University Hospital, Finland. Eligible patients were postmenopausal women (> 50 years old) with early-stage hormone receptor-positive BC treated with adjuvant letrozole for at least six months and developed symptoms of AV during this period. Exclusion criteria included premenopausal status, recent use of local estrogen therapy within the previous three months, irregular use of letrozole, and metastatic disease.

VVA diagnosis was based on patient-reported symptoms, with gynecologic examinations, including speculum examination with transvaginal sonography, performed for all participants at baseline. Vaginal Pap smears were used to determine the vaginal maturation index (VMI) by assessing the proportions of parabasal, intermediate and superficial cells in the vaginal wall, along with other cytological findings according to the Bethesda System for cervical cytology. Vaginal pH was measured using litmus paper placed on the vaginal wall until moistened, serving as an indicator of VVA.

Eligible patients were treated with Vagifem® (17β-estradiol hemihydrate) 10 μg vaginal tablets for 12 weeks. Patients were instructed to insert one vaginal tablet daily using the provided applicator for 14 consecutive days, followed by one tablet twice weekly (Monday and Thursday evenings). Blood samples were collected at baseline, prior to the initiation of study treatment, and at two, four, eight, and 12 weeks thereafter, within 24 to 60 hours of vaginal tablet administration. Serum was separated by centrifugation within 1 hour of collection and the samples were stored at -80°C until analysis.

Patients completed the EORTC QLQ-C30 and EORTC QLQ-BR23 questionnaires to assess QoL, with higher scores indicating better QoL or less QoL related symptoms, and the Women's Health Questionnaire (WHQ), where higher scores indicated greater distress and dysfunction, at baseline and after 12 weeks. Menopause-related symptoms were assessed using a structured 19-item questionnaire, while sexual function was evaluated with the McCoy Female Sexuality Questionnaire, which was completed by only half of the patients due to its limitation to sexually active participants. Higher scores on both questionnaires indicated greater severity or frequency of symptoms.

A follow-up gynecologic examination and oncology consultation were conducted at the end of the study to assess the patients' response to topical estradiol therapy. Patients who maintained serum E2 levels below LLOQ (< 5 pmol/L) and benefited from the therapy were considered for continued treatment off-study.

The primary objective was to analyze changes in serum E2 levels using two LC-MS/MS methods during concurrent adjuvant AI therapy and intravaginal estradiol treatment. Serum E2 levels were measured using both a routine LC-MS/MS method (Sciex Citrine™ Triple Quad™ LC-MS/MS system, E2-MS, HUSLAB, LLOQ 10 pmol/L) and a highly sensitive LC-MS/MS method (hsE2-MS, LLOQ 5 pmol/L, CV < 20%, LOD 1 pmol/L). The hsE2-MS method allowed for the detection of very low serum E2 concentrations, even below the LLOQ, within the range of 1-5 pmol/L, providing a precise assessment of the effect of letrozole and vaginal estrogen on E2 levels.

The intervention was considered unsuccessful if persistent elevation of E2 (> 5pmol/L in two consecutive tests) was observed after treatment initiation.

The local ethics committee of the Helsinki University Hospital approved the study protocol (No. 118). Informed consent was obtained from all participants included in the study. The trial was registered in the Helsinki and Uusimaa Hospital District Clinical Trials Register with EudraCT Number 2019-001234-34.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were postmenopausal women (> 50 years old) with early-stage hormone receptor-positive BC treated with adjuvant letrozole for at least six months and developed symptoms of AV during this period.

Exclusion Criteria:

* Exclusion criteria included premenopausal status, recent use of local estrogen therapy within the previous three months, irregular use of letrozole, and metastatic disease.

Min Age: 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 20 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Serum estradiol level | 12 weeks
  The primary objective was to analyze changes in serum E2 levels using two LC-MS/MS methods during concurrent adjuvant AI therapy and intravaginal estradiol treatment. ). Blood samples were collected at baseline, prior to the initiation of study treatment, and at two, four, eight, and 12 weeks thereafter, within 24 to 60 hours of vaginal tablet administration. Serum E2 levels were measured using both a routine LC-MS/MS method (Sciex Citrine™ Triple Quad™ LC-MS/MS system, E2-MS, HUSLAB, LLOQ 10 pmol/L) and a highly sensitive LC-MS/MS method (hsE2-MS, LLOQ 5 pmol/L, CV < 20%, LOD 1 pmol/L). The hsE2-MS method allowed for the detection of very low serum E2 concentrations, even below the LLOQ, within the range of 1-5 pmol/L, providing a precise assessment of the effect of letrozole and vaginal estrogen on E2 levels.

CONTACTS AND LOCATIONS:
Locations (1):
- HUS Comprehensive Cancer Center, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the current study are not publicly available due to the restrictions outlined in the consent form. However, they are available from the corresponding author on reasonable request.